CLINICAL TRIAL: NCT05481918
Title: Normalization of Gait After ACL Reconstruction: A Comparative Study Between Home-based Versus Standardized Therapy
Brief Title: Gait-based Evaluation of Early Rehabilitation After ACL Reconstruction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment problems
Sponsor: Karl Landsteiner University of Health Sciences (Other)
Collaborators: St. Pölten University of Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LSC18_018
Record Dates: First submitted 2022-06-20; First posted 2022-08-01 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2022-07

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: gait; exercise therapy; anterior cruciate ligament injuries; rehabilitation
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Investigator
Masking Description: A blinding of the patients is not possible, due to the nature of the study and the obviosity of group allocation. The principal investigator will be blinded to the allocation and will only get access to the coding list in special cases (e.g. harm). Furthermore, the principal investigator is not involved in the statistical analysis of data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standardized therapy (Active Comparator): The standardized outpatient rehabilitation program after ACL reconstruction contains 16 physiotherapeutic visits (groups+ individual), exclusively a stationary supervision.
  Therapies: stationary: 1x individual (30 min); from 2nd to 6th week: 2x individual (30 min), 5x group (30 min), 4x group (30min); From 6th week: 5x group (30 min)
  Interventions: Procedure: Standardized ambulant therapy after ACL reconstruction
- Home-based therapy (Experimental): The home-based program consists of five outpatient physiotherapeutic units (each 60 minutes) at the department of physical medicine and rehabilitation of the UHK. The timing of the physiotherapeutic supervisions was defined based on pre-existing studies, concerning home based therapy after ACL reconstruction. The five physiotherapeutic sessions will be executed by a physiotherapist in first, third, seventh, ninth and eleventh postsurgical week. In addition to a general information sheet, the patients of this group will receive phase-adapted training documents (with photographs) at each physiotherapeutic appointment.
  Interventions: Procedure: Home-based therapy after ACL reconstruction

INTERVENTIONS:
Procedure: Home-based therapy after ACL reconstruction — Five physiotherapeutic supervisions (individual) take place within the first 12-13 weeks after ACL reconstruction with focus on home exercises
  Arms: Home-based therapy
Procedure: Standardized ambulant therapy after ACL reconstruction — 16 physiotherapeutic supervisions (groups+ individual) take place within the first 12-13 weeks after ACL reconstruction.
  Arms: Standardized therapy

SUMMARY:
The objective of this study is to evaluate the regaining of a normal gait within the early rehabilitation (12-13 weeks postsurgical) after reconstruction of the anterior cruciate ligament (ACL). Therefore, two different rehabilitation programs (supervised versus home-based) will be compared.

A prospective, parallel-grouped trial with patients´ free choice of postsurgical therapy (home based versus supervised) will be conducted. One group will receive a well supervised, standardized rehabilitation program, while the other group will be instructed in a home-based rehabilitation program. Gait assessments will be carried out 6-7 weeks and 12-13 weeks postsurgical using standard 3D clinical gait analysis. Complementary, gait will also be evaluated using an Inertial Measurement Unit (IMU) three times postsurgical (6-7 weeks, 9-10 weeks, 12-13 weeks). Furthermore, various clinical parameters, like patient reported outcome measures (PROM), knee swelling, range of motion (ROM) will be taken presurgical as well as on days of gait assessment.

The study will show the impact of physiotherapeutic therapy on the early normalization of gait after ACL reconstruction. The results may help to build a better understanding of the required physiotherapeutic supervision after ACL surgery and if a home-based therapy can safely be recommended to specific patients.

DETAILED DESCRIPTION:
Design:

The study is designed as a prospective, parallel-grouped trial. The patient will have the free choice out of two postsurgical rehabilitation regimens. The baseline assessments will take place presurgical after the official enrolment procedure. After surgery, three follow ups are set (6-7, 9-10, 12-13 weeks postsurgical). 3D gait analysis will be performed on first and third series. Additionally, IMU gait analysis as well as the modified Star Excursion Balance Test (SEBT) will be performed . Furthermore, various clinical parameters, like patient reported outcome measures (PROM), knee swelling, range of motion (ROM) will be taken on assessment days.

Enrolment/Allocation/Blinding:

An appointment for checking eligibility will be made presurgical. If the patient is eligible, a signed informed consent will be collected and a continuous identification number will be defined by a central study coordinator. Further, the general personal data will be assessed, and presurgical measurements (e.g. ROM, knee swelling, PROM, height, weight) will be performed.

After surgery the patients can choose between a standardized rehabilitation program at the department of physical medicine and rehabilitation at University Hospital Krems (UHK) or a supervised home-based program.

A blinding of the patients is not possible, due to the nature of the study and the obviosity of group allocation. The principal investigator will be blinded to the allocation and will only get access to the coding list in special cases (e.g. harm). Furthermore, the principal investigator is not involved in the statistical analysis of data.

Rehabilitation programs:

Therapy Focus (both Groups):

Stationary setting: Reduction of swelling, gait training with crutches, introduction to a CPM (continuous passive motion) machine, instruction to exercises for home practice (active flexion and extension), stretching of ischiocrural muscles and M. iliopsoas From 2nd week postsurgical: Mobilisation of the patella, mobilisation of scars, gait training (beginning with partial weight-bearing), improvement of range of motion, progression of soft strengthening of knee flexion and extension.

From 6th week postsurgical: Focus on sensomotoric exercises. Progression of exercises for knee flexion and extension and intensified strengthening

Phase-adapted exercises for home-based Training:

Week 1-2:

1. Local cryotherapy (3x 20 min)
2. Mobilization of scars (after wound closure)
3. Active knee extension in supine position
4. Active knee extension in supine position with padding underneath the heel
5. Active knee extension in prone position
6. Active knee flexion and extension in closed chain in supine position (heel contact with floor)
7. Activating of M. quadriceps femoris and ischiocrural muscles by tensing

Week 3-6:

1. Local cryotherapy (3x 20 min) after exercise, if required
2. Active knee extension in supine position without padding
3. Progression: full knee extension while standing/half seated
4. Active knee extension in supine position with padding underneath the heel
5. Active knee extension in supine position in open chain (no floor contact of the foot)- max. 20° flexion
6. Knee flexion and extension in closed chain in supine position (heel contact to the floor), with TheraBand
7. Activating M. quadriceps and ischiocrural muscles with foot-support on the wall in

   * 30° knee-flexed position/ 60-90° knee-flexed position
8. Mini-Squats (holding on a chair back)
9. Bridging- extending the knee, while lying supine with raised pelvic
10. Raising the operated leg lying in lateral position with extended knee/ with flexed knee
11. Knee extension and load takeover without crutches in standing Position

Week 7-8:

1. Local cryotherapy (3x 20 min) after exercise, if required
2. Active knee extension in supine position with padding underneath the heel
3. Active knee extension in supine position in open chain (no floor contact of the foot)- max. 20° flexion
4. Active knee flexion and extension in closed chain in supine position (progression: with gymnastic ball)
5. Activating M. quadriceps and ischiocrural muscles with foot-support on the wall (or to progress on gymnastic ball) in 30° knee-flexed position/ 90° knee-flexed position
6. Knee extension and flexion in seated position in closed chain. Extension against resistance of TheraBand
7. Squats (30°-0° flexion/ 80°-60° flexion)
8. Bridging- extending both knees alternately, while lying supine with raised pelvic
9. Extension of knee and hip in lateral position (on healthy side) with contact of injured limb with the wall
10. Standing on one foot
11. Walking frontwards and backwards with active extended knees

Week 9-10:

1. Local cryotherapy (3x 20 min) after exercise, if required
2. Active knee extension in supine position with padding underneath the heel
3. Active knee flexion and extension in closed chain in supine position
4. Knee extension and flexion in seated position in closed chain (heel contact with floor) with eyes closed. Extension against resistance of TheraBand.
5. Squat lunges to the side. The knees are alternately flexed, while the toes of the contralateral limb tip the floor to the side.
6. Bridging- extending both knees alternately, while lying supine with raised pelvic
7. Standing on one foot, while the other knee is flexed 90° and the foot pushes against a wall behind
8. Standing on one foot, doing different exercises with the upper body (e.g. arm movement, head rotation)
9. Walking frontwards and backwards with active extended knees
10. Planking on forearms (exercise time increases)

Week 11-12:

1. Cryotherapy, if required
2. Active knee flexion and extension in closed chain in supine position
3. Variation of Squats (eyes closed, arm movement, full knee ROM, stabilizing in 60°/90° flexion)
4. Variation of Squat lunges to the side (eyes closed, arm movement, rotation of upper body, stabilizing in 90° flexion)
5. Lunges moving forward
6. Standing on one foot, ankles connected with TheraBand. Moving free limb back and to the side against resistance of TheraBand. Difficulty increases with different arm tasks or closed eyes.
7. Standing on one foot, doing different exercises with the upper body (e.g. arm movement, head rotation)
8. Variation of lunges
9. Stride leaps
10. Planking on forearms

Independently of group allocation, each patient is offered a prescription of an electrotherapeutic device (Schuhfried Company, Vienna, Austria) with two electrodes (8x12cm) for quadriceps muscle strengthening with surge current for home application.

Training diaries:

Patients of both rehabilitation programs will be encouraged to keep training diaries to monitor progression in load increase, repetitions of exercises and frequency in the period of home training. Additional treatments shall also be documented (e.g. surge current). The diaries between the groups differ, as the standard-group will receive only one general sheet to document their training for the whole study period, while the home-based group will receive an extra sheet for every phase (5 documents), where all exercises can be selected separately.

Ethical aspects:

All participants will be informed about the nature and the scope of the study and will give a written consent. The trial has been registered and received an ethical approval of the Committee for Scientific Integrity and Ethics of the Karl Landsteiner University Krems. The registration number is 1038/2019. Participants may withdraw from the study anytime, without giving a specific reason. Furthermore, if a participant may take obvious physiological harm by staying within the study protocol, the principal investigator can decide to remove him/her from the study.

Sample size calculation and statistical procedures:

For the statistical analysis a matched pair t-test will be used. The matching criteria will be the Tegner score (maximum one point difference) and the age of the participants (maximum five years difference).

The required number of patients was calculated beforehand using the software nQuery version 8.5. The sample size estimation is based on the primary outcome parameter (step length symmetry) after a literature review. According to the calculation 24 pairs are needed to detect a statistical effect size of 0.6 with a power of 80 percent. Considering the usual drop-out rates and the impossibility of finding matching partners, for estimated a third of the participants, the sample size was set with 45 persons per group.

ELIGIBILITY:
Inclusion Criteria:

* Surgery at University Hospital Krems (UHK), Austria
* Age 18-60 years
* Surgery-timing less than six months posttraumatic
* Isolated ACL rupture with or without small concomitant injuries

Exclusion Criteria:

* Relevant concomitant injuries of the musculoskeletal system
* Old injuries of the lower limbs, which influence the normal gait pattern (including ACL re-ruptures)
* Relevant orthopaedic pre-existing conditions, especially of the lower limbs.
* Severe internistic and neurological concomitant diseases, which have an impact on the cardiorespiratory fitness or the physiologic gait
* Patients who do not speak or understand the German or English language properly

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Changes in step length | 6-7 and 12-13 weeks after ACL reconstruction
  The primary outcome will be the regaining of a symmetrical step length in 3D gait analysis. Therefor, the symmetry index by Robinson et al. will be used. Data will be collected using a motion capture system (VICON, Oxford, UK), comprising of 12 infrared-cameras at a sampling rate of 150 Hz A full body marker set with a total of 50 retro-reflective spherical markers with a diameter of 14 mm and 9 mm will be attached bilaterally on each participant using double-sided tape. Markers will be placed at bony landmarks according to the manual of the Cleveland Clinic Marker Set and the Plug in Gait model (upper extremity). The 3D marker trajectories of all markers will be reconstructed and processed using the VICON Nexus analysis software (v. 2.5, Oxford, UK). Kinetic data will be collected simultaneously by using three force plates (AMTI, Watertown, USA) at a sampling rate of 1500 Hz.

SECONDARY OUTCOMES:
Kinetic gait parameters (3D gait analysis) | 6-7 and 12-13 weeks after ACL reconstruction
  Unit: Nm/kg Kinetic gait parameters, which are known to be altered after ACL reconstruction will be analyzed. Known alterations of kinetic parameters of the knee are the maximum moment of flexion, extension, adduction and external rotation. Concerning the hip, alterations of the maximum moment of extension and flexion are common.
  The 3D gait analysis system is described in Outcome 1.
Kinematic gait parameters (3D gait analysis) | 6-7 and 12-13 weeks after ACL reconstruction
  Unit: degrees. Kinematic gait parameters, which are known to be altered after ACL reconstruction will be analyzed. Known altered kinematic parameters of the knee are the maximum adduction, flexion, internal and external tibial rotation. For the hip, the known altered parameters are the maximum flexion and adduction, are described.
  The 3D gait analysis system is described in Outcome 1.
Step length (IMU) | 6-7, 9-10, 12-13 weeks after ACL reconstruction
  Unit: centimeter. Distance from the heel of one foot-strike to the heel of the opposite foot-strike The used system (BTS Bioengineering Corp., Quincy, USA) includes an IMU (BTS G-Sensor 2) with a triaxial accelerometer (multiple sensitivities from 2-16g), a triaxial gyroscope (multiple sensitivities form 250 - 2000°/s, 16bit/axes) and a triaxial magnetometer (1200T, 13bit).
Kinematic pelvic parameters (IMU) | 6-7, 9-10, 12-13 weeks after ACL reconstruction
  Unit: degrees. All three dimensions of pelvic movement are measured (anterior and posterior tilt in sagittal plane; depression and elevation in frontal plane; rotation in transversal plane;) The system used is described in Outcome 4.
Temporal gait parameters (3D+IMU) | 6-7, 9-10, 12-13 weeks after ACL reconstruction
  Unit: seconds. Parameters included are Stance Time and Swing Time. The systems used are described in Outcome 1. and 4.
Range of Motion (knee) | Presurgical, 6-7, 9-10, 12-13 weeks after ACL reconstruction
  The testing of the knee ROM will be performed according to the neutral zero method (flexion/extension) with a digital, long axis goniometer (30x30cm)
Knee circumference | Presurgical, 6-7, 9-10, 12-13 weeks after ACL reconstruction
  The circumference of the knee will be measured on three locations on the extended leg (5 centimeter proximal the upper patella pole/ height of joint gap/ height of fibular head).
Modified Star Excursion Balance Test (mSEBT) | 12-13 weeks postsurgical
  The modified SEBT is used to assess the knee stability in the anterior, the posteromedial and the posterolateral direction after injury. Therefore, three strips of tape will be placed on the laboratory floor, forming an ypsilon. For the assessment the participants stand on one leg in the intersection area of the strips. Three attempts are performed for each leg with the aim to achieve maximal reach of the non-stance limb in the directions, marked by the strips.
Modified Lysholm Score | Presurgical, 6-7, 9-10, 12-13 weeks after ACL reconstruction
  These questionnaire is commonly used in clinical and scientific fields to assess the function, symptoms and the level of daily activity in patients after knee injury or with knee pain.
  Max. points are 100 (=best outcome)
International Knee Documentation Committee Subjective Knee Form (IKDC) | Presurgical, 6-7, 9-10, 12-13 weeks after ACL reconstruction
  This questionnaire is commonly used in clinical and scientific fields to assess the function, symptoms and the level of daily activity in patients after knee injury or with knee pain.
  Max. points are 87 (=100%)
Tegner activity score | Presurgical and 12-13 weeks after ACL reconstruction
  These questionnaire is commonly used in clinical and scientific fields to obtain the score of activity level in patients with knee disorders. It complements other functional scores like the Lysholm Score.
  Max. points are 10 (=best activity)
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Presurgical, 6-7, 9-10, 12-13 weeks after ACL reconstruction
  This questionnaire is commonly used in clinical and scientific fields to assess the function, symptoms and the level of daily activity in patients after knee injury or with knee pain.
  Max. points are 168 (=100%).

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Ernst, Dr., Principal Investigator — Karl Landsteiner University of Health Sciences
Locations (3):
- Austria (3):
  - Department of Biomechanics, Karl Landsteiner University of Health Sciences, Krems, Lower Austria
  - Department of Physical Medicine and Rehabilitation, University Hospital Krems., Krems, Lower Austria
  - Institute of Health Sciences, Department of Health, St. Pölten University of Applied Sciences, Sankt Pölten, Lower Austria